CLINICAL TRIAL: NCT00002029
Title: Long-Term Nutritional Support in Patients With the Acquired Immunodeficiency Syndrome: Comparison of Liposyn III 2 Percent With Liposyn II 20 Percent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 041A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Weight Loss; Parenteral Nutrition, Total; AIDS-Related Opportunistic Infections; Liposyn; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Weight Loss; Hyperphagia; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: Fat Emulsion 2%
Drug: Fat Emulsion 20%

SUMMARY:
To compare two lipid emulsions in the long-term parenteral alimentation of patients with AIDS in relation to: Clinical effectiveness. Effect on immunologic function. Effect on HIV load as measured by p24 antigen levels. Effect on relative HIV infectivity.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* All drugs used for the standard treatment of opportunistic infections.
* Other drugs used for the treatment of other AIDS conditions if they have been started more than 3 months prior to study entry.

Patients must have:

* Diagnosis of AIDS.
* Weight loss of > 10 percent premorbid body weight.
* Presenting diagnosis of either opportunistic infection or Kaposi's sarcoma.
* Require home total parenteral nutrition (TPN) for a period of approximately 3 months.
* Life expectancy = or > 90 days.

Prior Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Life expectancy < 90 days.
* Biliary stasis.
* History of drug abuse.

Patients with the following are excluded:

* Life expectancy < 90 days.
* Biliary stasis.
* History of drug abuse.

Prior Medication:

Excluded within 3 months of study entry:

* Immunomodulators.
* Experimental antiviral DT. History of drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Intracare Inc, Miami, Florida
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey

REFERENCES:
- [Background] Singer P, Rubinstein A, Askanazi J, Calvelli T, Lazarus T, Kirvela O, Katz DP. Clinical and immunologic effects of lipid-based parenteral nutrition in AIDS. JPEN J Parenter Enteral Nutr. 1992 Mar-Apr;16(2):165-7. doi: 10.1177/0148607192016002165. PMID 1556814